CLINICAL TRIAL: NCT06399120
Title: Diagnostic Performance of Endocytoscopy for Colorectal Lesions
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Hong Xu, Director, Head of Gastroenterology and Endoscopy Center, Principal Investigator, Clinical Professor, The First Hospital of Jilin University
Other Study IDs: 24K102-001
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Lesions
Keywords: endocytoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer is the third most common malignancy worldwide and the second leading cause of cancer-related death. About 70% of colorectal cancers develop through the adenoma-cancer pathway. Early detection and resection of colorectal neoplastic lesions significantly reduce the morbidity and mortality of colorectal cancers. Colonoscopy is considered to be the preferred method for screening for colorectal lesions. However, as the number of endoscopic resection increases, the costs associated with pathological diagnosis of endoscopic resection and resection specimens increase year by year. In clinical practice, it will be very important and urgent to correctly judge the nature of colorectal lesions to avoid pathological diagnosis and then realize optical biopsy. Therefore, to clarify the endoscopic diagnosis of colorectal lesions, many endoscopic techniques have been applied clinically. Such as narrow-band imaging, magnifying narrow-band imaging endoscopy, magnifying chromoendoscopy and endocytoscopy. Endocytoscopy has two modes, EC-NBI mode and EC-staining mode. EC-NBI mode is to observe the microvessel on the mucosal surface of colorectal mucosa after switching the endoscopy to NBI mode. EC-V pattern is used to observe microvessels and then endoscopic diagnosis is performed. The EC-staining mode was that the cell nuclei and glandular duct morphology of colorectal lesions could be observed by endocytoscopy after chemical staining. Endocytoscopic diagnosis is performed clinically after observation of glandular ducts and nuclei. However, current studies on the diagnostic value of endoscopy in colorectal lesions are all retrospective studies with small samples, and there is a lack of clinical studies based on chinese population. Therefore, our center intends to conduct a study of a large sample to explore the diagnostic value of endoscopy in colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* colorectal lesions

Exclusion Criteria:

* non-epithelial tumors
* a history of inflammatory bowel disease
* lesions without clear EC images
* specific pathological types
* familial adenomatous polyposis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators analyzed only endoscopically or surgically resected colorectal lesions that had been observed and diagnosed with endoscopic methods by endoscopists that were ultimately performed histopathologic examination.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
sensitivity of diagnosing colorectal lesions using endocytoscopy | May 2025
  The percentage of patients with a specific type of colorectal disease who received a positive result by endocytoscopy.
specificity of diagnosing colorectal lesions using endocytoscopy | May 2025
  The percentage of patients with non-specific types of colorectal disease who received a negative result using endocytoscopy.
accuracy of diagnosing colorectal lesions using endocytoscopy | May 2025
  The percentage of correct results that is obtained by endocytoscopy.
positive predictive value of diagnosing colorectal lesions using endocytoscopy | May 2025
  The percentage of patients with positive results when using endocytoscopy to diagnose colorectal lesions.
negative predictive value of diagnosing colorectal lesions using endocytoscopy | May 2025
  The percentage of non-patients with negative results when using endocytoscopy to diagnose colorectal lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Mingqing Liu, Changchun, Jilin, China